CLINICAL TRIAL: NCT01291329
Title: Phase 2 Study of Intracoronary Human Wharton's Jelly- Derived Mesenchymal Stem Cells (WJ-MSCs) Transfer in Patients With ST-segment Elevation Acute Myocardial Infarction (AMI)
Brief Title: Intracoronary Human Wharton's Jelly- Derived Mesenchymal Stem Cells (WJ-MSCs) Transfer in Patients With Acute Myocardial Infarction (AMI)
Acronym: WJ-MSC-AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Collaborators: Chinese PLA General Hospital (Other); General Hospital of Chinese Armed Police Forces (Other); First People's Hospital of Foshan (Other)
Responsible Party: Lian Ru Gao, Cardiology Division of Navy General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006AA02Z469
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: stem cell; acute ST-Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WJ-MSC (Experimental): Wharton's jelly- Derived Mesenchymal Stem Cells Transfer
  Interventions: Genetic: intracoronary human umbilical WJ-MSC transfer

INTERVENTIONS:
Genetic: intracoronary human umbilical WJ-MSC transfer — intracoronary infusion of WJ-MSCs or placebo medium into the infarct artery 4-7 days after successful reperfusion therapy.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of intracoronary human umbilical Wharton's jelly-derived mesenchymal stem cell (WJ-MSC) transfer in patients with ST-segment elevation acute myocardial infarction.

DETAILED DESCRIPTION:
It has been demonstrated that MSCs have the potential to differentiate into cardiomyocytes both in vitro and in vivo. Several clinical trials have been performed using autologous bone marrow-derived MSCs, but the results of these trials have been unsatisfactory because of a low number of MSCs in older patients and in those with coronary heart disease. WJ-MSCs from the human umbilical cord matrix which are of epiblastic origin and contain both human embryonic stem cell (hESC) and human mesenchymal stem cell markers appear to have a number of important advantages: they do not raise ethical issues, are widely multipotent, are not tumorigenic, and are not immunogenetic. Because of a short population doubling time they can be rapidly scaled up in large numbers. We performed a double-blind, placebo-controlled, multicenter trial, randomly assigning 160 patients with acute ST-segment elevation myocardial infarction to receive an intracoronary infusion of WJ-MSCs or placebo medium into the infarct artery 4-7 days after successful reperfusion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years of age；
2. Patients with 1st acute ST-elevation myocardial infarction (AMI) who undergo successful primary percutaneous coronary intervention (PCI) thrombolysis in myocardial infarction (TIMI) flow grade 3, but have a substantial residual left ventricular regional wall-motion abnormality measured by 2-D echocardiography.
3. No contraindications to undergoing cell-therapy procedure within 1 weeks after AMI and PCI.
4. Hemodynamic stability-defined as no requirement for intra-aortic balloon pump or for inotropic or blood-pressure supporting medications.
5. Consent to protocol and agree to comply with all follow-up visits and studies.

Exclusion Criteria:

1. Presence of cardiogenic shock ( defined as systolic blood pressure < 80 mmHg requiring intravenous pressors or intra-aortic balloon counterpulsation);
2. Major bleeding requiring blood transfusion after acute reperfusion treatment;
3. A history of leucopenia;
4. Thrombocytopenia;
5. Hepatic or renal dysfunction;
6. Evidence for malignant diseases;
7. Unwillingness to participate;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Quantify myocardium metabolic and perfusion measured by F-18-fluorodeoxyglucose (F-18-FDG) postremission tomography (PET) and 99 mTctetrofosmine single-photon (SPET), as well as global left ventricular ejection fraction measured by echocardiography. | 4 months- 1 year
  The primary endpoints were differences between the two treatments and from baseline to 4 months in quantitative myocardial metabolic and perfusion images, as measured by 18F-FDG positron emission tomography and 99 mTctetrofosmine single-photon imaging. Left ventricular ejection fraction is measured by 16-segment 2-D echocardiography.

SECONDARY OUTCOMES:
Secondary endpoints: safety will be determined by the assessment of major adverse coronary events (MACE). | 4 months-1year
  Safety will be determined by the assessment of major adverse coronary events (MACE) defined as cardiac death, peri-procedural myocardial infarction, or any repeat coronary intervention at 4 months-1year. Furthermore, safety is also determined by the occurrence of stent thrombosis, arrhythmias events. immune system disorders. The trial will be monitored by a Data and Safety Monitoring Board (DSMB) and the trial will be discontinued in case of safety concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Ru Gao, MD, Study Chair — Cardiology Division of Navy General Hospital
Locations (1):
- Fu Cheng Lu 6, Beijing, China

REFERENCES:
- [Result] 1.Monya Baker. How to fix a broken heart? Nature. 2009; 460:18-19. 2.Psaltis PJ, Zannettino A, Worthley SG. Mesenchymal stromal cells potential for cardiovascular repair. Stem cells.2008; 10:1634. 3.Deryl L, Mark LT, Weiss, et al. Concise review : wharton's jelly-derived cells are a primitive stromal cell population. Stem Cells. 2008 ; 26 :591-599. 4.Nekanti U, Rao VB, Bahirvani AG, Ta M, et al. Long-term Expansion and Pluripotent Marker Array Analysis of Wharton's Jelly-Derived Mesenchymal Stem Cells. Stem Cells and Dev. 2010; 19:117-130. 5.Chen MY, Lie PC, Li ZL. Endothelial differentiation of Wharton's jelly-derived mesenchymal stem cells in comparison with bone marrow-derived mesenchymal stem cells. Exp Hematol. 2009;37(5):629-40.. 6.Wu KH, Mo XM, Zhou, B. et al. Cardiac potential of stem cells from whole human umbilical cord tissue. Journal of Cellular Biochemistry. 2009; 107:926-932.
- [Derived] Gao LR, Chen Y, Zhang NK, Yang XL, Liu HL, Wang ZG, Yan XY, Wang Y, Zhu ZM, Li TC, Wang LH, Chen HY, Chen YD, Huang CL, Qu P, Yao C, Wang B, Chen GH, Wang ZM, Xu ZY, Bai J, Lu D, Shen YH, Guo F, Liu MY, Yang Y, Ding YC, Yang Y, Tian HT, Ding QA, Li LN, Yang XC, Hu X. Intracoronary infusion of Wharton's jelly-derived mesenchymal stem cells in acute myocardial infarction: double-blind, randomized controlled trial. BMC Med. 2015 Jul 10;13:162. doi: 10.1186/s12916-015-0399-z. PMID 26162993